CLINICAL TRIAL: NCT03030495
Title: IMaging and Physiologic Predictors of Atherosclerotic Progression in Deferred Lesions With Contemporary Medical Treatment Based on Fractional Flow Reserve-guided Strategy
Brief Title: Registry of Comprehensive Imaging and Physiological Evaluation of Deferred Lesions Based on FFR
Acronym: IMPACT-FFR
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Inje University Ilsan Paik Hospital (Other); Ulsan University Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Other Study IDs: IMPACT16453143
Record Dates: First submitted 2016-12-20; First posted 2017-01-25 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Ischemic Heart Disease
Keywords: Ischemic Heart Disease; Stable angina; Fractional flow reserve; Index of Microcirculatory Resistance; Coronary Flow Reserve; Intravascular Imaging
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Overt microvascular disease: Fractional flow reserve>0.80, coronary flow reserve<2 & Index of microvascular resistance>25U
  Interventions: Device: Comprehensive physiologic evaluation; Device: Intravascular imaging devices
- No Overt microvascular disease: Fractional flow reserve>0.80, coronary flow reserve>2 & Index of microvascular resistance<25U
  Interventions: Device: Comprehensive physiologic evaluation; Device: Intravascular imaging devices

INTERVENTIONS:
Device: Comprehensive physiologic evaluation — Comprehensive physiologic evaluation using pressure-temperature sensor wire to measure fractional flow reserve, coronary flow reserve, index of microcirculatory resistance
  Other Names: Comprehensive physiologic evaluation using pressure-temperature sensor wire
Device: Intravascular imaging devices — Intravascular ultrasound or optical coherence tomography
  Other Names: Intravascular ultrasound or optical coherence tomography

SUMMARY:
1. To compare the risk of atherosclerotic lesion progression and subsequent patient-oriented composite outcomes (all-cause mortality, any MI, or any Ischemia-driven repeat revascularization) between deferred lesions with or without over microvascular disease, defined as physiological classification
2. To explore independent predictors of atherosclerotic lesion progression in deferred lesions based on fractional flow reserve-guided strategy and treated by contemporary medical treatment

DETAILED DESCRIPTION:
The coronary artery system has 3 components with different functions: conductive epicardial coronary arteries, arterioles, and capillaries. When any one of these systems fails, myocardial ischemia can occur. Therefore, the presence of epicardial coronary artery stenosis is not necessarily a prerequisite for ischemic heart disease (IHD). Although it has not been established that microvascular disease is independent of macrovascular disease, clinical studies have consistently shown that the presence of microvascular disease is an independent predictor of poor clinical outcomes, especially in patients with acute myocardial infarction (MI).

The pressure-derived fractional flow reserve (FFR) index has become a standard invasive method to evaluate the functional significance of epicardial coronary artery stenosis, and clinical outcomes of FFR-guided percutaneous coronary intervention (PCI) have proven to be better than those of angiography-guided PCI or medical treatment. Although FFR-guided PCI has been reported to improve patient outcomes and FFR is now regarded as the gold-standard invasive method to assess the functional significance of coronary artery stenosis, there is still room for further improvement in the diagnosis and treatment of patients with high FFR. In the FAME II study, 14.6% of the registry arm (FFR > 0.80 and deferral of PCI) experienced persistent angina, and 9.0% of these patients had clinical events during a 2-year follow-up period.

Therefore, microvascular assessment using coronary flow reserve (CFR) and the index of microcirculatory resistance (IMR) can provide additional diagnostic and prognostic insights for IHD patients, especially in those with high FFR.

Recently, Lee et al. (JACC 2016) investigated clinical outcomes among patients with high-FFR and deferred revascularization, according to physiologic classification using CFR and IMR. Lee et al. firstly presented that 7.0% of patients with high FFR had high IMR and low CFR and were regarded as having overt microvascular disease. Although the proportion of patients with high FFR who had overt microvascular disease was small, Group D had the poorest clinical outcomes during follow-up. The presence of overt microvascular disease was an independent prognostic factor in patients with high FFR. In addition, the presence of overt microvascular disease had additive prognostic value aside from clinical risk factors, with significantly improved discriminant function of the prediction model. These results suggest that the invasive physiologic assessment for microvascular disease combined with CFR and IMR can help identify patients at high risk for future cardiovascular events among those with high FFR.

Previous studies have shown that the presence of microvascular disease is associated with a higher risk of cardiovascular events such as cardiac death, MI, or revascularization in patients without flow-limiting epicardial stenosis. Several mechanisms have been proposed for the association of microvascular disease and poor clinical outcomes. In addition to myocardial ischemia, microvascular disease is reported to be associated with endothelial dysfunction and inflammatory activity that precedes intimal thickening, lipid deposition in the macrovascular system, and coronary vasomotor dysfunction. In a study by Dhawan et al., coronary microvascular dysfunction in patients with non-obstructive coronary artery disease was associated with higher serum high-sensitivity C-reactive protein and a higher frequency of thin-cap fibroatheroma.

In the Lee et al.'s study, the higher clinical event rates in patients with overt microvascular disease resulted from cardiac death and revascularization rates higher than those of the other groups. These results imply that the presence of overt microvascular disease can induce accentuated atherosclerotic progression and subsequent clinical events including cardiac death and ischemia-driven repeat revascularization.

Therefore, the IMaging and Physiologic Predictors of Atherosclerotic Progression in Deferred Lesions with Contemporary Medical Treatment based on Fractional Flow Reserve-guided Strategy (IMPACT-FFR registry) was designed to compare the risk of atherosclerotic plaque progression and subsequent clinical events between deferred lesions with or without over microvascular disease, defined as physiological classification and also to explore independent predictors of atherosclerotic lesion progression in deferred lesions based on fractional flow reserve-guided strategy and treated by contemporary medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years
* Patients suspected with ischemic heart disease
* Patients with intermediate degree of stenosis (30-70% stenosis by visual estimation) with fractional flow reserve of >0.80 in major epicardial coronary artery amenable to stent implantation or vessel size≥2.5 mm
* Patients whose coronary stenosis were evaluated by invasive imaging techniques (intravascular ultrasound and optical coherence tomography) and physiologic assessment (coronary flow reserve, index of microcirculatory resistance, and fractional flow reserve)
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic or imaging evaluation and he/she or his/her legally authorized representative provides written informed consent to any study related procedure

Exclusion Criteria:

* End-staged renal disease on peritoneal dialysis or hemodialysis (estimated GFR < 15mL/min)
* Acute hepatic injury
* Cardiogenic shock (systolic blood pressure < 90mmHg or requiring inotropics to maintain blood pressure > 90mmHg)
* The patient has a known hypersensitivity or contraindication to any of the following medications: statin, ezetimibe, heparin, aspirin, clopidogrel, prasugrel, ticagrelor
* Non-cardiac co-morbid conditions are present with life expectancy <2 year (per site investigator's medical judgment)
* Unable to perform invasive imaging study (intravascular ultrasound and optical coherence tomography) or physiologic assessment (coronary flow reserve, index of microcirculatory resistance, and fractional flow reserve)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate degree of stenosis (30-70% stenosis by visual estimation) with fractional flow reserve of >0.80 in major epicardial coronary artery amenable to stent implantation or vessel size ≥2.5 mm.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
patient-oriented composite outcome | 24 months
  a composite of all-cause death, MI, any repeat revascularization

SECONDARY OUTCOMES:
patient-oriented composite outcome | 12 months
  a composite of all-cause death, MI, any repeat revascularization
patient-oriented composite outcome | 60 months
  a composite of all-cause death, MI, any repeat revascularization
All-cause death | 24 months
  All-cause death
cardiac death | 24 months
  cardiac death
Target-vessel nonfatal MI | 24 months
  Target-vessel nonfatal MI
Non-target vessel nonfatal MI | 24 months
  Non-target vessel nonfatal MI
All-cause nonfatal MI | 24 months
  All-cause nonfatal MI
Seattle Angina Questionnaires | 24 months
  Angina severity measured with Seattle Angina Questionnaires
Change in normalized total atheroma volume | 12 months
  TAVnormalized = [Σ (EEM CSA - lumen CSA) / no. of images in pullback images in cohort] X median no. of images in cohort
Change in total atheroma volume index | 12 months
  Indexed total atheroma volume (TAVi): Σ(EEM CSA -lumen CSA)/plaque length
Change in fibrous cap thickness by OCT | 12 months
  Change in fibrous cap thickness by OCT at 12-month
Change in Plaque burden at minimum lumen area site | 12 months
  Change in Plaque burden at minimum lumen area site at 12-month Plaque burden = (EEM-MLA)/EEM x 100
Change in Fractional flow reserve | 12 months
  Change in Fractional flow reserve at 12-month
Change in coronary flow reserve | 12 months
  Change in coronary flow reserve at 12-month
Change in index of microcirculatory resistance | 12 months
  Change in index of microcirculatory resistance at 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center; Bon-Kwon Koo, MD, PhD, Study Chair — Seoul National University Hospital; Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center; Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (4):
- South Korea (4):
  - Keimyung University Dongsan Medical Center, Daegu
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked